CLINICAL TRIAL: NCT02680015
Title: Understanding the Effects of Intervention on the Brain in Autism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Marquette University (Other)
Responsible Party: Principal Investigator, Amy Vaughan Van Hecke, Professor of Psychology, Marquette University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HR 2020
Record Dates: First submitted 2016-02-04; First posted 2016-02-11 (Estimated); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Autism Spectrum Disorder; Asperger Disorder; PDD-NOS; Autism
Keywords: PEERS; friendships; brain
MeSH Terms: conditions — Autism Spectrum Disorder; Asperger Syndrome; Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): Immediate enrollment in the PEERS group.
  Interventions: Behavioral: PEERS
- Waitlist Group (No Intervention): Research measures while waiting for PEERS; will receive PEERS within one year.

INTERVENTIONS:
Behavioral: PEERS — Social-behavioral intervention designed to help individuals with Autism Spectrum Disorder make and keep friends.
  Other Names: Program for the Education and Enrichment of Relational Skills
  Arms: Experimental Group

SUMMARY:
This study examines how the PEERS (Laugeson & Frankel, 2010; Laugeson, 2016) social-behavioral intervention affects social relationships and brain development and function in autistic preschoolers, adolescents, and young adults.

ELIGIBILITY:
Inclusion Criteria:

* Verbal, speaking in full sentences
* Meets ASD criteria
* Meets IQ criteria >70

Exclusion Criteria:

* schizophrenia or bipolar disorder

Ages: 4 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2010-08; Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Social Responsiveness Scale (SRS: Constantino, 2005) | within two weeks of PEERS completion
  Questionnaire completed by caregivers on social function and autism symptoms. Will be aggregated by group; no individual reports will be used.
Test of Adolescent Social SKills (TASSK: Laugeson & Frankel, 2010) | within two weeks of PEERS completion
  Questionnaire completed by participants with Autism Spectrum Disorder. Measures knowledge of the PEERS intervention concepts. Will be aggregated by group; no individual reports will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Van Hecke, PhD, Principal Investigator — Marquette University
Locations (1):
- Marquette University, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No